CLINICAL TRIAL: NCT07329192
Title: First Required Medical Examination of the Newborn After Discharge From the Maternity Hospital: Does the Choice of a General Practitioner Facilitate Its Completion Within the Recommended Timeframe ?
Brief Title: Study on How Parents' Anticipated Choice of a Doctor at the Maternity Hospital Influences the Newborn's First Post-discharge Consultation
Acronym: GENS2-VIE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0045
Record Dates: First submitted 2025-12-08; First posted 2026-01-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Newborn Infant; Newborn
Keywords: infant; newborn; postnatal care (MeSH); general practitioner; physician; primary care; pediatric primary care; Post-discharge Follow-up; Health Services Accessibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newborn: newborn
  Interventions: Other: Advance Selection of a General Practitioner

INTERVENTIONS:
Other: Advance Selection of a General Practitioner — This exposure refers to parents selecting a general practitioner for their newborn before discharge from the maternity hospital.
  It represents a routine-care organizational choice that may influence whether the first post-discharge medical examination is completed within the recommended period. No study-specific procedures or treatments are administered.

SUMMARY:
The goal of this observational study is to determine whether, in a population of well-informed parents, choosing a general practitioner at the maternity hospital facilitates the completion of the newborn's first required medical examination within the second week of life.

The main question it aims to answer is: Does selecting a general practitioner before leaving the maternity hospital allow the newborn's first medical examination to be completed within the recommended period?

Participants will be asked to complete an initial questionnaire, which will be given to them before leaving the maternity hospital, and then a second questionnaire by telephone one month later.

DETAILED DESCRIPTION:
For eligible newborns, an information sheet will be provided to the parents or legal guardians.

Parents or legal guardians who have been informed of the study and do not object to their child's participation will receive a questionnaire between the second postnatal day (D2) and discharge from the maternity ward.

Each completed questionnaire will be collected prior to discharge. The research team will then contact the parents by telephone on day 30 (±3 days) to administer the second questionnaire and record their responses.

ELIGIBILITY:
Inclusion Criteria:

* Term newborn ≥ 37 weeks of gestation
* Birth weight > 3000 g
* Growth > 5th percentile according to Fenton curves
* No diagnosed or suspected pathology during antenatal care or the maternity stay
* No postnatal complications requiring temporary hospitalization in the neonatal unit or kangaroo care unit

Exclusion Criteria:

* Pathology diagnosed or suspected in the newborn during the maternity hospital stay.
* Requirement for temporary hospitalization in a neonatal unit or kangaroo care unit, including but not limited to: neonatal jaundice, abnormal oxygenation or laboratory findings, suspected early-onset bacterial infection, transient respiratory distress requiring more than 2 hours of non-invasive ventilation at birth, monitoring of mother-infant bonding, or maternal treatments during pregnancy necessitating clinical monitoring.
* Language barrier in both parents.
* Parents (legal guardians) informed of the study and having declined participation for themselves and their child.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy term newborns recruited prior to discharge from the maternity hospital. Included infants are healthy term newborns (≥37 weeks of gestation, birth weight >3000 g) with no antenatal or postnatal pathology requiring hospitalization. Parents or legal guardians must understand the study information and not object to participation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Timely completion of the newborn's first post-discharge medical examination | at 1 month
  Assessment of whether the newborn's first medical examination after discharge from the maternity hospital is performed within the recommended period (second week of life, between day 8 and day 15).
  The outcome is measured as a binary variable: completed within the recommended period / not completed within the recommended period.

SECONDARY OUTCOMES:
Sociodemographic data of the parents' choice of physician for the newborn's first consultation | at day 0
  Assessment of parental (sociodemographic, organizational, informational) and neonatal (clinical, perinatal) characteristics associated with the selection of the physician designated to perform the newborn's first post-discharge consultation.
Questions regarding the first post-hospitalization consultation | at maternity (assessed up to day 7)
  Evaluation of the information received by parents and their level of knowledge regarding the purpose, timing, and importance of the newborn's first post-discharge consultation, including awareness of recommended guidelines.
Concordance between the physician designated in maternity and the physician who performed the consultation | at 1 month
  Comparison between the physician chosen by parents before hospital discharge and the physician who actually performed the newborn's first medical examination.
Factors associated with delayed completion of the newborn's first consultation | at 1 month
  Identification of parental, organizational, and neonatal factors associated with completion of the first consultation after the recommended period.
  Outcome measured as timely vs. delayed, with analysis of associated covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Marion BATHANY, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No